CLINICAL TRIAL: NCT06643143
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of IkT-001Pro in Pulmonary Arterial Hypertension
Brief Title: A Phase 2 Study of IkT-001Pro in Pulmonary Arterial Hypertension (PAH)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has undergone sponsorship and design changes.
Sponsor: Inhibikase Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IkT-001Pro-702
Record Dates: First submitted 2024-10-09; First posted 2024-10-16 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Arterial Hypertension (PAH); Pulmonary Arterial Hypertension (PAH) (WHO Group 1 PH)
Keywords: Pulmonary Arterial Hypertension; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo Control (Experimental): Placebo
  Interventions: Drug: Placebo
- 300mg (Experimental): 300mg
  Interventions: Drug: IkT-001Pro
- 500mg (Experimental): 500mg
  Interventions: Drug: IkT-001Pro

INTERVENTIONS:
Drug: IkT-001Pro — IkT-001Pro
  Arms: 300mg; 500mg
Drug: Placebo — Placebo
  Arms: Placebo Control

SUMMARY:
This is a randomized, double-blind, multi-center, placebo-controlled dose-ranging clinical trial of two IkT-001Pro doses in patients with PAH designed to assess safety, tolerability and efficacy. It will enroll approximately 150 participants at up to 50 sites globally. The study consists of two parts, a 26 week placebo controlled treatment period (Part A) followed by a 36 month extension period (Part B).

DETAILED DESCRIPTION:
This is a randomized, double-blind, multi-center, placebo-controlled dose-ranging clinical trial of two IkT-001Pro doses in patients with PAH. This study will enroll approximately 150 participants at up to 50 sites globally.

The study consists of two parts, a 26 week placebo controlled treatment period (Part A) followed by a 36 month extension period (Part B). Those participants that pass the screening process will be randomized during the baseline visit to either the low dose (300mg) or placebo in a 2:1 ratio.

After two weeks participants will return to the clinic; upon confirmation that the participants are tolerating their dose, those that are on active treatment will be randomized to either 300mg or 500mg active treatment arms in a 1:1 manner. Those participants on placebo will remain on placebo for the rest of the 26-week placebo controlled treatment period. The final randomization structure for the 26-week placebo controlled treatment period will be such that participants are randomized in a 1:1:1 scheme to the 300 mg, 500 mg or placebo groups.

Participants who have not discontinued early will transition to a 36 month extension period. Participants who transition to the extension period will remain on the dose that they were assigned to after the two week acclimation period. Participants who were randomized to the placebo group will be re-randomized 1:1 to either the 300mg or 500mg IkT-001Pro treatment groups. The study will be unblinded and investigators will be given treatment assignments once the primary endpoint analysis is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 70 years of age (inclusive) at the time of signing the informed consent.
2. Capable of giving signed ICF.
3. Documented diagnostic right heart catheterization (RHC) at any time prior to screening confirming the diagnosis of WHO PAH Group 1 in any of the following subtypes:

   1. Idiopathic PAH
   2. Heritable PAH
   3. Drug/toxin-induced PAH
   4. PAH associated with CTD
   5. PAH associated with simple, congenital systemic-to-pulmonary shunts at least 1 year following repair
4. Symptomatic PH classified as WHO FC II or III
5. Baseline RHC performed during the Screening Period documenting a minimum PVR of

   ≥ 400 dyn.sec.cm-5 (≥5 WU) and a pulmonary capillary wedge pressure (PCWP) or left ventricular end-diastolic pressure of ≤ 15 mmHg.

   a. NOTE: At least 50% of study population needs to have PVR ≥ 800 dyn.sec.cm-5.
6. On stable doses of background PAH therapy (i.e., patient-specific dose goal for each therapy already achieved) for at least 90 days prior to screening; for infusion prostacyclins, dose adjustment within 10% of optimal dose is allowed per medical practice.

   a. For those taking sotatercept their dosing regimen should be stable for at least 6 months prior to screening
7. 6MWD ≥ 150 and ≤ 500 m repeated twice at screening (measured at least 4 hours apart, but no longer than 1 week), and both values are within 15% of each other (calculated from the highest value).

Exclusion Criteria:

1. Diagnosis of PAH WHO Groups 2, 3, 4, or 5
2. Diagnosis of the following PAH Group 1 subtypes: human immunodeficiency virus (HIV)-associated PAH and PAH associated with portal hypertension. Exclusions in PAH Group 1 should also include schistosomiasis-associated PAH and pulmonary veno-occlusive disease
3. Uncontrolled systemic hypertension as evidenced by sitting systolic BP > 160 mmHg or sitting diastolic BP > 100 mmHg during screening visit after a period of rest
4. Personal or family history of long QT syndrome (LQTS) or sudden cardiac death
5. Pulmonary function tests (PFT) completed no more than 24 weeks before the screening period (or completed at the Screening Visit). Following criteria must are considered exclusionary
6. Cerebrovascular accident within 3 months prior to the screening visit
7. Currently receiving moderate or strong Cytochrome P450 (CYP) 3A4/5 inducers or CYP3A4/5 inhibitors (except for topical administration)
8. Currently receiving or anticipated need to receive anticoagulants
9. Currently receiving or anticipated need to receive more than one anti-platelet medication. The use of prostacyclins is not considered exclusionary. Note that sotatercept is not considered anti-platelet therapy
10. Initiation of an exercise program for cardiopulmonary rehabilitation within 90 days prior to the screening visit or planned initiation during the study (participants who are stable in the maintenance phase of a program and who will continue for the duration of the study are eligible)
11. History of atrial septostomy within 180 days prior to the screening visit
12. Current participation in another investigational clinical trial and/or receipt of any investigational medication within 90 days prior to screening
13. Estimated glomerular filtration rate (eGFR) < 30 mL/min/m2 (as defined by the Modification of Diet in Renal Disease [MDRD] equation)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect on PVR in participants with WHO functional class II-III PAH treated with IkT-001Pro compare to placebo | Through study completion, an average of 26 weeks with 36 months of extension
  Change in PVR at 26 weeks compared to baseline
To assess the safety and tolerability of two IkT-001Pro doses in PAH | Through study completion, an average of 26 weeks with 36 months of extension
  Incidence and temporal profile of treatment-emergent adverse events (TEAEs) evaluated by type/nature, severity/intensity, seriousness, and relationship to study intervention

SECONDARY OUTCOMES:
To characterize the effects of two IkT-001Pro doses on symptoms and characterics of Pulmonary Arterial Hypertension | Through study completion, an average of 26 weeks with 36 months of extension
  Change from Baseline to Week 26 in 6 minute walk test.
To characterize the effects of two IkT-001Pro doses on symptoms and characterics of Pulmonary Arterial Hypertension | Through study completion, an average of 26 weeks with 36 months of extension
  Time to death or the first occurrence of any of the following clinical worsening events; Lung or heart-lung transplantation, Atrial septostomy, Hospitalization for worsening of PAH (≥ 24 hours) or Deterioration of PAH defined by both of the following events occurring at any time, even if they began at different times, as compared to their baseline values.
To characterize the effects of two IkT-001Pro doses on symptoms and characterics of Pulmonary Arterial Hypertension | Through study completion, an average of 26 weeks with 36 months of extension
  Number of participants who improve in WHO FC or who maintain or achieve a low risk score at Week 26 versus baseline using the ESC/ERS 4-strata model.
To assess the PK of IkT-001Pro in participants with PAH | Through study completion, an average of 26 weeks with 36 months of extension
  PK parameters of IkT-001Pro
Part B : To assess the long-term safety and tolerability of two IkT-001Pro doses in PAH | Through study completion, an average of 26 weeks with 36 months of extension
  Incidence and temporal profile of treatment-emergent adverse events (TEAEs) evaluated by type/nature, severity/intensity, seriousness, and relationship to study intervention
To characterize the effects of two IkT-001Pro doses on symptoms and characterics of Pulmonary Arterial Hypertension | Through study completion, an average of 26 weeks with 36 months of extension
  Change from Baseline to Week 26 in the Physical Impacts domain score of Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT®)
To characterize the effects of two IkT-001Pro doses on symptoms and characterics of Pulmonary Arterial Hypertension | Through study completion, an average of 26 weeks with 36 months of extension
  Change from Baseline to Week 26 in the Cardiopulmonary Symptoms domain score of Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT®)
To characterize the effects of two IkT-001Pro doses on symptoms and characterics of Pulmonary Arterial Hypertension | Through study completion, an average of 26 weeks with 36 months of extension
  Change from Baseline to Week 26 in the Cognitive/Emotional Impacts domain score of Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT®)